CLINICAL TRIAL: NCT00395421
Title: A Partially-blinded, Randomized, Parallel-group Study to Evaluate the Potential Pharmacokinetic and Pharmacodynamic Interactions Between Valopicitabine and Ribavirin When Administered in Combination With Pegylated Interferon Alfa-2a in Treatment-naive Patients With Chronic Hepatitis C
Brief Title: Study to Evaluate Drug-drug Interaction Between Valopicitabine and Ribavirin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: John Z. Sullivan-Bólyai, MD, MPH, Idenix Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NV-08A-008
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Hepatitis C
Keywords: treatment-naive
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — valopicitabine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): NM283(200 mg QD)plus Peg-IFNα-2a (180 µg QW)
  Interventions: Drug: NM283 plus Peg-IFNα-2a

INTERVENTIONS:
Drug: NM283 plus Peg-IFNα-2a — 200 mg QD 180 µg QW

SUMMARY:
This study is being conducted to see if the investigational medication, valopicitabine, is safe to use in combination with ribavirin, a drug approved by the FDA for treating hepatitis C infection.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical history compatible with chronic hepatitis C and compensated liver disease
* Has not previously received anti-viral therapy for hepatitis C infection

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient is co-infected with hepatitis B virus and/or HIV

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Atlanta, Georgia
  - Fairfax, Virginia